CLINICAL TRIAL: NCT01024335
Title: Dronabinol Naltrexone Treatment for Opioid Dependence
Acronym: Domino
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, National Institute on Drug Abuse (NIDA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: #5962 DA027124; R01DA027124 (NIH); DPMC (Other: NIDA)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2014-09-05 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Opioid Dependence
Keywords: opioid dependence; naltrexone; vivitrol; dronabinol; marinol
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Dronabinol; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone and placebo (Active Comparator): A long-acting, injectable form of naltrexone 380 mg (Vivitrol) will be administered once per month while placebo will be taken daily for the first 5 weeks of treatment.
  Interventions: Drug: Naltrexone and placebo
- Naltrexone and dronabinol (Experimental): A long-acting, injectable form of naltrexone 380 mg (Vivitrol) will be administered once per month (the total of two injections, once at the end of hospitalization, and once at end of first month of outpatient treatment), while dronabinol (15 mg bid) will be taken daily for the first 5 weeks of treatment.
  Interventions: Drug: injectable naltrexone and dronabinol

INTERVENTIONS:
Drug: injectable naltrexone and dronabinol — Injectable form of naltrexone 380 mg (Vivitrol) will be administered once per month plus dronabinol 15 mg bid for the first 5 weeks of treatment.
  Arms: Naltrexone and dronabinol
Drug: Naltrexone and placebo — Injectable form of naltrexone 380 mg (Vivitrol) will be administered once per month plus placebo bid for 5 weeks.
  Arms: Naltrexone and placebo

SUMMARY:
The goal of this two-year study is to test the efficacy of dronabinol as an adjunct to maintenance treatment with naltrexone in opioid-dependent individuals. We hypothesize that administering dronabinol during detoxification and during the first few weeks of naltrexone treatment will lead to improved naltrexone tolerability, resulting in better naltrexone compliance and treatment retention, and ultimately a reduction in opioid use and relapse rates.

DETAILED DESCRIPTION:
The goal of this two-year study is to test the efficacy of dronabinol as an adjunct to maintenance treatment with naltrexone in opioid-dependent individuals. We are proposing a randomized, double-blind, placebo controlled, parallel-groups, 8 week study of relapse prevention in opioid-dependent individuals. Participants will be randomized into one of two conditions (1) Naltrexone and Placebo (N=20) and (2) Naltrexone and dronabinol 15 mg bid (N=40). Treatment will be delivered in an outpatient setting except for the initial phase of inpatient detoxification, lasting 8 days. A long-acting, injectable form of naltrexone 380 mg (Vivitrol) will be administered once per month (the total of two injections), while dronabinol or placebo will be taken daily. In addition, patients will receive a psychosocial intervention that will include elements of motivational interviewing and cognitive-behavioral relapse prevention therapy. The primary aim is to test the efficacy of dronabinol in improving tolerability of naltrexone induction and reducing attrition during detoxification and the first two months of naltrexone treatment. The primary outcome will be the severity of opiate withdrawal and craving. The secondary outcome will be will be retention in treatment at study's end.

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult, aged 18-60.
* 2. Meets Diagnostic and Statistical Manual -IV criteria for current opiate dependence disorder of at least six months duration, supported by a positive urine for opiates and a positive naloxone challenge test if the diagnosis is unclear.
* 3. Have a history of marijuana use (more than 30 occasions lifetime)
* 4. Voluntarily seeking treatment for opioid dependence
* 5. In otherwise good health based on complete medical history, physical examination, vital signs measurement, ECG, and laboratory tests (hematology, blood chemistry, urinalysis) within normal ranges.
* 6. Able to give informed consent.

Exclusion Criteria:

* 1. Physiologically dependent on alcohol or sedative-hypnotics with impending withdrawal.
* 2. Patients meeting current criteria for cannabis abuse or dependence, and those who used cannabis in the week prior to study entry as documented by the positive toxicology
* 3. Current Diagnostic and Statistical Manual -IV criteria of other substance use disorders. Exceptions include cannabis abuse or dependence, nicotine dependence, cocaine abuse or dependence, alcohol abuse or alcohol dependence without physiological dependence as long as opioid dependence is a primary disorder. Alcohol dependence with physiological dependence is exclusionary.
* 4. Significant current suicidal risk or 1 or more suicide attempts within the past year
* 5. History of accidental drug overdose in the last three years defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.
* 6. Positive serum pregnancy test, lactation, or unwillingness to use a satisfactory method of birth control
* 7. Active psychiatric disorder which might interfere with participation or make participation hazardous, including Diagnostic and Statistical Manual -IV organic mental disorder, psychotic disorder, or bipolar disorder with mania
* 8. History of allergic reaction, adverse reaction, or sensitivity to any study medication.
* 9. Acute hepatitis with serum glutamic-oxaloacetic transaminase or serum glutamic-pyruvic transaminase > 3 times the upper end of the laboratory normal range (chronic hepatitis is acceptable as we have found naltrexone treatment well tolerate and safe among patients with chronic hepatitis)
* 10. Currently prescribed or regularly taking opiates for chronic pain or medical illness.
* 11. Current participation in a methadone maintenance treatment program and/or regular use of illicit methadone (>30 mg per week).
* 12. Current participation in another intensive psychotherapy or substance abuse treatment program or participation in another treatment study.
* 13. Concurrent treatment with psychotropic medications

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone and Placebo | Naltrexone and Dronabinol
Started | 20 | 40
Completed | 7 | 14
Not Completed | 13 | 26

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone and Placebo | Naltrexone and Dronabinol | Total
Number analyzed (Participants) | 20 | 40 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (11.1) | 38.5 (11.6) | 38.1 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 16 | 34 | 50
Race/Ethnicity, Customized [Number; unit: participants]
  White | 12 | 23 | 35
  Black | 2 | 3 | 5
  Hispanic | 5 | 13 | 18
  Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Opiate Withdrawal Measured by the Subjective Opiate Withdrawal Scale (SOWS) .
Description: The Subjective Opiate Withdrawal Scale is a self-administered 16 scale containing 16 symptoms ranging in severity from 0 (not at all) to 4 (extremely). The SOWS total score is the sum of 16 items, ranging from 0 (no opiate withdrawal ) to 64 ( severe opiate withdrawal). Values from multiple assessments during the 8-week outpatient phase were averaged.
Time Frame: 3x/week during 8 weeks of the trial or study participation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Naltrexone and Placebo | Naltrexone and Dronabinol
Number analyzed (Participants) | 20 | 40
units on a scale | 11.16 (6.13) | 13.36 (10.55)

2. Primary Outcome: Retention
Description: Of those participants randomized to the naltrexone and dronabinol arm, the number that completed all 8 weeks of treatment.
Time Frame: retention over 8 weeks.
Measure: Number; unit: participants
Arm/Group | Naltrexone and Placebo | Naltrexone and Dronabinol
Number analyzed (Participants) | 20 | 40
participants | 7 | 14

ADVERSE EVENTS:
Arm/Group | Naltrexone and Placebo | Naltrexone and Dronabinol
Serious Adverse Events (participants affected / at risk) | 2/20 | 1/40
Other Adverse Events (participants affected / at risk) | 10/20 | 28/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone and Placebo (N=20) | Naltrexone and Dronabinol (N=40)
Pruritis and facial swelling (General disorders) | 0 (0) | 1 (1) — A participant in the dronabinol treatment arm developed symptoms of pruritis and facial swelling two days after receiving an injection of naltrexone. A dermatologist determined that the rash was most likely not related to the study medication.
Dehydration (General disorders) | 1 (1) | 0 (0) — One participant in the placebo arm was hospitalized for symptoms of dehydration during the first week of the outpatient phase.
Kidney infection and dislocated arm (General disorders) | 1 (1) | 0 (0) — A participant in the placebo arm was hospitalized for treatment of a kidney infection and dislocated arm, which occurred 3 weeks after discontinuation of study participation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone and Placebo (N=20) | Naltrexone and Dronabinol (N=40)
Insomnia (Psychiatric disorders) | 7 (7) | 17 (17)
Mood changes (Psychiatric disorders) | 4 (4) | 5 (5)
Increased/decreased appetite (General disorders) | 2 (2) | 2 (2)
Nausea/vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 7 (7)
Headache (General disorders) | 2 (2) | 3 (3)
Body Aches (General disorders) | 1 (1) | 3 (3)
GI Distress (Gastrointestinal disorders) | 3 (3) | 4 (4)
Sweating/chills (General disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No